CLINICAL TRIAL: NCT04600921
Title: Ertugliflozin to Reduce Arrhythmic Burden in Implantable Cardioverter-defibrillators (ICD)/Cardiac Resynchronisation Therapy(CRT) patientS (ERASe-Trial) - a Phase III Study
Brief Title: Ertugliflozin to Reduce Arrhythmic Burden in ICD/CRT patientS (ERASe-Trial) - a Phase III Study
Acronym: ERASE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The feasibility (recruitment) of the high number of patients (402 patients with HFrEF or HFmrEF) was impossible due to the rapid increase in SGLT2 inhibitors in patients with heart failure.
Sponsor: Medical University of Graz (Other)
Collaborators: Klinikum Klagenfurt am Wörthersee (Other); Elisabethinen Hospital (Other); Medical University Innsbruck (Other); Medical University of Vienna (Other); General Hospital Linz (Other); Landesklinkum Wiener Neustadt (Other); Klinik Ottakring (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DvL-2020-01
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Heart Failure With Mid Range Ejection Fraction; Implantable Cardioverter-Defibrillators; Cardiac Resynchronization Therapy
Keywords: Ertugliflozin; Sodium dependent glucose transporter-2 inhibitor (SGLT-2); Heart failure; ICD; CRT; ventricular tachycardia (VT)
MeSH Terms: conditions — Heart Failure; Tachycardia, Ventricular | interventions — ertugliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ertugliflozin (Active Comparator): The subject will receive Ertugliflozin 5mg.
  Interventions: Drug: Ertugliflozin 5 mg
- Placebo (Placebo Comparator): The subject will receive Placebo 5mg.
  Interventions: Drug: Placebo 5mg

INTERVENTIONS:
Drug: Ertugliflozin 5 mg — The subject will receive Ertugliflozin 5mg orally once daily for 52 weeks.
  Other Names: Steglatro
  Arms: Ertugliflozin
Drug: Placebo 5mg — The subject will receive Placebo 5mg orally daily for 52 weeks.
  Other Names: Sugar pills
  Arms: Placebo

SUMMARY:
The recent study is planned to investigate the impact of Ertugliflozin on total burden of ventricular arrhythmias. Further objectives will be number of therapeutic interventions of implanted devices, atrial fibrillation, heart failure biomarker and changes in physical function quality of life, stress and anxiety.

DETAILED DESCRIPTION:
This is a randomized, double-blind (patients and physicians), placebo controlled multi-center study to evaluate the effect of ertugliflozin 5mg once daily (p.o.) for 52 weeks on the ventricular arrhythmic burden and markers of physical and mental well-being as well as biomarker for Heart Failure with reduced Ejection Fraction (HFrEF) and heart failure with mid-range ejection fraction (HFmrEF) patients with ICD±CRT therapy. The study will be conducted in 8 experienced sites in Austria with an aim to enrol 402 patients to evaluate the overall study hypothesis.

Therefore, three study visits will be carried out (baseline, 1-year follow-up visit and a telephone visit 4 weeks after visit 2). As part of the two on-site study visits, study-specific measures, a blood sample and an echocardiographic examination will be performed. The trial is completed by a telephone visit 4 weeks after the second on-site visit (week 52).

It is anticipated that the study will run for 30 months.

ELIGIBILITY:
Inclusion Criteria:

1. HFrEF or HFmrEF, and ICD±CRT therapy > 3 months
2. at least 10 documented VT episodes (either nsVT (non-sustained ventricular tachycardia) or sVT (sustained ventricular tachycardia) ± ICD (mplantable cardioverter-defibrillator) treatment) within the last 12 months plus:

   * nt-proBNP > 500pg/mL or
   * Left-ventricular Ejection Fraction (LV-EF) < 35% or
   * hospitalization for heart failure within the last 12 months or
   * > 100 nsVTs within the last 12 months
   * > 1 sVT/VF (ventricular function) within the last 12 months
3. Informed consent has to be given in written form.
4. estimated glomerular filtration rate (eGFR) > 30 ml/min/1.73m2
5. Blood pressure before first drug dosing: blood pressure systolic > 100 mmHg
6. Blood pressure before first drug dosing: blood pressure diastolic > 60 mmHg

Exclusion Criteria:

1. Any other form of diabetes mellitus than type 2 diabetes mellitus, history of diabetic ketoacidosis
2. Ongoing ventricular arrhythmia
3. Known allergy to SGLT-2 inhibitors
4. Haemodynamic instability as defined by intravenous administration of catecholamine, calciumsensitizers or phosphodiesterase inhibitors
5. >1 episode of severe hypoglycemia within the last 6 months under treatment with insulin or sulfonylurea
6. Planned catheter ablation for ventricular arrhythmia
7. Planned explantation of ICD, or planned up/downgrade to/from CRT-D device
8. Existing therapy with SGLT-2 inhibitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk von Lewinski, Assoc-Prof., Principal Investigator — Medical University of Graz
Locations (8):
- Austria (8):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt, Carinthia
  - Kepler Universitätsklinikum Linz, Linz, Upper Austria
  - Medical University of Graz, Graz
  - Universitätsklinikum Innsbruck, Innsbruck
  - Ordensklinikum Linz Elisabethinen, Linz
  - Medizinische Universität Wien, AKH Wien, Vienna
  - Wilhelminenspital, Vienna
  - Landesklinikum Wiener Neustadt, Wiener Neustadt

REFERENCES:
- [Derived] Benedikt M, Oulhaj A, Rohrer U, Manninger M, Tripolt NJ, Pferschy PN, Aziz F, Wallner M, Kolesnik E, Gwechenberger M, Martinek M, Nurnberg M, Roithinger FX, Steinwender C, Widkal J, Leiter S, Zirlik A, Stuhlinger M, Scherr D, Sourij H, von Lewinski D. Ertugliflozin to Reduce Arrhythmic Burden in Patients with ICDs/CRT-Ds. NEJM Evid. 2024 Oct;3(10):EVIDoa2400147. doi: 10.1056/EVIDoa2400147. Epub 2024 Sep 1. PMID 39217453
- [Derived] von Lewinski D, Tripolt NJ, Sourij H, Pferschy PN, Oulhaj A, Alber H, Gwechenberger M, Martinek M, Seidl S, Moertl D, Nurnberg M, Roithinger FX, Steinwender C, Stuhlinger M, Zirlik A, Benedikt M, Kolesnik E, Wallner M, Rohrer U, Manninger M, Scherr D; ERASe study group. Ertugliflozin to reduce arrhythmic burden in ICD/CRT patients (ERASe-trial) - A phase III study. Am Heart J. 2022 Apr;246:152-160. doi: 10.1016/j.ahj.2022.01.008. Epub 2022 Jan 16. PMID 35045327

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ertugliflozin | Placebo
Started | 25 | 30
Completed | 22 | 24
Not Completed | 3 | 6
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: The subject will receive Placebo 5mg.
  Placebo 5mg: The subject will receive Placebo 5mg orally once daily for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Ertugliflozin | Placebo | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] — The inclusion criteria for age was 18 to 80 years.
  years | 65 (11) | 66 (12) | 65 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 20 | 22 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 24 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 22 | 24 | 46
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — Height was meausred at the screening visit. Weight was measured at all visits. BMI was calculated using the formula as follows: BMI = weight (kg) / height² (m²)
  kg/m² | 28.6 (5.3) | 28.2 (6.3) | 28.4 (5.8)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Systolic blood pressure was meausred in sitting position at all visits.
  mmHg | 136 (13) | 131 (21) | 133 (18)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Diastolic blood pressure was measured in sitting position at all visits.
  mmHg | 87 (12) | 81 (15) | 84 (14)
Heart rate [Mean (Standard Deviation); unit: beats/minute] — Heart rate was recorded at all visits after resting for 5 minutes in a sitting position.
  beats/minute | 68 (12) | 72 (13) | 70 (13)
Baseline medications [Count of Participants; unit: Participants]
  Angiotensin-converting enzyme inhibitor/ Angiotensin receptor blocker | 13 | 12 | 25
  Beta-blockers | 18 | 21 | 39
  Mineralocorticoid receptor blocker | 12 | 14 | 26
  Angiotensin receptor blocker and neprilysin inhibitor | 6 | 8 | 14
  Loop diuretics | 9 | 15 | 24
  Dihydropyridine (CCB) | 2 | 2 | 4
  Verapamil/Diltiazem (CCB) | 0 | 0 | 0
  Digitalis | 2 | 2 | 4
  Amiodarone/sotalol | 4 | 6 | 10
  Supplemental Magnesium | 6 | 5 | 11
  Platelet aggregation inhibitors | 4 | 6 | 10
  Anticoagulants | 15 | 12 | 27
  Statins | 14 | 15 | 29
Baseline arrhythmic burden, 12 months prior [Mean (Standard Deviation); unit: Number of episodes]
  Sustained ventricular tachycardia or Ventricular fibrillation | 19 (44) | 6 (10) | 12 (32)
  Non-sustained Ventricular tachycardia episodes | 22 (33) | 27 (57) | 25 (47)
Left ventricular ejection fraction, 12 months prior [Mean (Standard Deviation); unit: percentage] | 36 (8) | 38 (14) | 37 (11)
Potassium concentration [Mean (Standard Deviation); unit: mmol/l] | 4.5 (0.6) | 4.5 (0.50) | 4.5 (0.5)
Magnesium concentration [Mean (Standard Deviation); unit: mmol/l] | 0.9 (0.1) | 0.8 (0.1) | 0.9 (0.1)
C-reactive protein level [Mean (Standard Deviation); unit: mg/l] | 3 (3) | 2 (2) | 2 (3)
Estimated glomerular filtration rate [Mean (Standard Deviation); unit: ml/min/1.73m²] | 65 (21) | 57 (16) | 61 (18)
NTproBNP levels [Mean (Standard Deviation); unit: ng/l] | 1141 (1598) | 2370 (2714) | 1782 (2311)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Supraventricular Tachycardia (svT)/ Ventricular Fibrillation (VF) Episodes
Description: Change in number of supraventricular tachycardia (svT)/ ventricular fibrillation (VF) episodes from baseline to week 52
Time Frame: 52 weeks
Population: We randomized 55 patients, 25 in the ertugliflozin group and 30 in the placebo group. 5 patients from the placebo group and 3 from the placebo group withdrew consent before termination of the trial. 1 patient from the placebo group died without sufficient telemetric data. Consequently, only 46 patients were analysed including 22 in the ertugliflozin group and 24 in the placebo group.
Measure: Mean (Standard Deviation); unit: Number of episode
Arm/Group | Ertugliflozin | Placebo
Number analyzed (Participants) | 22 | 24
Number of episode | 3 (6) | 13 (34)
Statistical Analysis 1: Comparison: Ertugliflozin vs Placebo; We compared the rate of sVT/VF episodes between experimental arms after 52 weeks.The initial sample calculation was based on the mathematical formula provided by Zhu and Lakkis for comparing event rates of two negative binomial distributiuons. To detect a 30% reduction in VT/VF episode rates in the ertugliflozin group compared to placebo group, with 80% power and an alpha level of 0.05, accounting for 5% drop out in each group, a total sample size of 402 was estimated to be required; Test type: Superiority — The parameters required to calculate sample size were the expected rate of VT/VF episodes/year in the placebo group, the minimal VT/VF rate ratio to be detected in the ertugliflozin group compared with the placebo group, the average follow-up of treatment duration, the negative binomial dispersion parameter, type 1 error probability, and the desired power; p < 0.001, Negative binomial regression model — The yearly rate ratio was adjusted for baseline number of sVT/VF episodes; A prespecified sensitivity analysis was done to mitigate the effect of outliers by using the robust estimation approaches for negative binomial model; Rate Ratio = 0.16, 95% CI 2-sided [0.04 to 0.61] — Ertugliflozin is the numerator and the placebo is the denominator

2. Secondary Outcome: Number of Nonsustained Ventricular Tachycardia (nsVT) Episodes
Description: Number of nonsustained ventricular tachycardia (nsVT) episodes from baseline to week 52
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: Number of episodes
Arm/Group | Ertugliflozin | Placebo
Number analyzed (Participants) | 22 | 24
Number of episodes | 28 (54) | 130 (322)
Statistical Analysis 1: Comparison: Ertugliflozin vs Placebo; The number of incident nsVT episodes were analyzed using a beta binomial model; Test type: Superiority; Rate Ratio = 0.34, 95% CI 2-sided [0.12 to 0.97]

3. Secondary Outcome: Number of Episodes of Appropriate Implantable Cardioverter-defibrillator Therapies
Description: Number of episodes of appropriate Implantable cardioverter-defibrillator therapies from baseline to week 52.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: Number of ICD therapies
Arm/Group | Ertugliflozin | Placebo
Number analyzed (Participants) | 22 | 24
Number of ICD therapies | 5 (8) | 10 (33)
Statistical Analysis 1: Comparison: Ertugliflozin vs Placebo; The number of appropriate ICD therapies were analyzed by using beta binomial model; Test type: Superiority; Rate Ratio = 0.47, 95% CI 2-sided [0.13 to 1.81]

4. Secondary Outcome: Change in NTproBNP Levels
Description: Change in NTproBNP levels from baseline to week 52
Time Frame: 52 weeks
Measure: Median (Inter-Quartile Range); unit: ng/l
Arm/Group | Ertugliflozin | Placebo
Number analyzed (Participants) | 22 | 24
ng/l | 143 [-6 to 300] | 101 [-103 to 322]
Statistical Analysis 1: Comparison: Ertugliflozin vs Placebo; The change in NTproBNP levels was analyzed by using a multiple linear regression model; Test type: Superiority; p > 0.05, Regression, Linear; Difference in mean change = 0.17, 95% CI 2-sided [-0.35 to 0.69]

5. Secondary Outcome: Change in HbA1c Levels
Description: Change in HbA1c levels from baseline to week 52
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Ertugliflozin | Placebo
Number analyzed (Participants) | 22 | 24
mmol/mol | -0.9 (5.1) | -1.33 (4.9)
Statistical Analysis 1: Comparison: Ertugliflozin vs Placebo; The change in HbA1c levels from baseline to week 52 was analyzed by multiple linear regression model; Test type: Superiority; Mean Difference (Final Values) = 0.72, 95% CI 2-sided [-1.69 to 3.13]

6. Secondary Outcome: Number of Hospitalizations
Description: Number of hospitalizations from baseline to week 56
Time Frame: 56 weeks
Measure: Mean (Standard Deviation); unit: number of hospitalizations
Arm/Group | Ertugliflozin | Placebo
Number analyzed (Participants) | 22 | 24
number of hospitalizations | 0.7 (1.0) | 1.3 (2.2)
Statistical Analysis 1: Comparison: Ertugliflozin vs Placebo; Test type: Superiority; Rate Ratio = 0.6, 95% CI 2-sided [0.2 to 1.7]

7. Secondary Outcome: Atleast One Hospitalization Due to Heart Failure
Description: It is the number of patients with at least one hospital re-admission due to heart failure from baseline to 56 weeks
Time Frame: 56 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ertugliflozin | Placebo
Number analyzed (Participants) | 22 | 24
Participants | 1 | 4

8. Secondary Outcome: Number of Hospitalizations Due to Heart Failure
Description: It is the number of hospital re-admissions due to heart failure from baseline to 56 weeks.
Time Frame: 56 weeks
Measure: Number; unit: Number of patients
Arm/Group | Ertugliflozin | Placebo
Number analyzed (Participants) | 22 | 24
Number of patients | 1 | 12

9. Secondary Outcome: Duration of Hospital Stay
Description: It is the number of days of hospital stay from baseline to 56 weeks
Time Frame: 56 weeks
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Ertugliflozin | Placebo
Number analyzed (Participants) | 22 | 24
Number of days | 3.6 (5.3) | 10.4 (23.5)

10. Secondary Outcome: Cardiovascular Mortality
Description: Difference in Cardiovascular mortality between treatment groups from randomisation to week 56
Time Frame: 56 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ertugliflozin | Placebo
Number analyzed (Participants) | 22 | 24
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events are recorded from baseline to 56 weeks
Arm/Group | Ertugliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 3/25 | 3/30
Serious Adverse Events (participants affected / at risk) | 10/25 | 21/30
Other Adverse Events (participants affected / at risk) | 4/25 | 2/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin (N=25) | Placebo (N=30)
Hospitalization due to cardiovascular event (Cardiac disorders) | 3 (5) | 4 (5)
Cardiovascular death (Cardiac disorders) | 1 | 2
Hospitalization due to non-cardiovascular causes (General disorders) | 2 (2) | 7 (9)
Non-cardiovascular death (General disorders) | 2 | 1
Infectious disease (Infections and infestations) | 1 (1) | 3 (3)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Any Hospitalization (General disorders) | 10 (12) | 21 (33)
Death (General disorders) | 3 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin (N=25) | Placebo (N=30)
Hepatic Injury (Hepatobiliary disorders) | 0 | 0 — Adverse event of special interest
Renal Injury (General disorders) | 0 | 1 — Adverse event of special interest
Metabolic acidosis and diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 — Adverse event of special interest
Event involving lower limb amputation (Musculoskeletal and connective tissue disorders) | 0 | 0 — Adverse event of special interest
Urinary tract infection (Infections and infestations) | 1 (1) | 0 — Other adverse event
Genital fungal infection (Infections and infestations) | 1 (6) | 1 (4) — Other adverse event
Hypotension (Blood and lymphatic system disorders) | 1 (1) | 0 — Other adverse event
Polyuria (General disorders) | 1 (1) | 0 — Other adverse event
Total Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 — Other adverse event

LIMITATIONS AND CAVEATS:
An important limitation is the lack of generalizability because our study predominantly included White men. A second limitation is that our trial was prematurely stopped, and thus we did not achieve the planned power to accurately assess our primary end point. In addition, seven patients withdrew their consent to continue in the trial. Therefore, the results of our primary and key secondary end points must be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT04600921/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT04600921/SAP_001.pdf